CLINICAL TRIAL: NCT02292953
Title: Variation in Serum Prolactin Levels in Response to Ovum Pickup for Patients Undergoing ICSI & it's Effect on Pregnancy Rate
Brief Title: Variation in Serum Prolactin Levels During IntraCytoplasmic Sperm Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed M.Kamel, Lecturer of Obstetric & Gynecology, Kasr El Aini Hospital
Other Study IDs: A13952014
Record Dates: First submitted 2014-11-10; First posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Infertility
Keywords: ICSI; Ovum Pickup; Embryo Transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Serum Prolactin levels — blood samples will be drawn from patients undergoing ICSI to analyse serum prolactin levels

SUMMARY:
The purpose of the study is to determine whether or not stressful conditions such as ovum pick and awaiting Embryo Transfer is associated with significant increase in serum Prolactin (PRL) concentration in some normo-prolactinemic patients undergoing intracytoplasmatic sperm injection (ICSI) & possible effect on implantation & pregnancy rate.

DETAILED DESCRIPTION:
Methodology in details:

After applying inclusion and exclusion criteria to infertile patients scheduled for start of ICSI cycle at kasr alainy assisted reproduction unit, and taking the patient's informed consent for all blood samples that will be drawn from her.

The baseline serum prolactin level is recorded and the first blood sample is scheduled to be taken in operating room just before induction of anesthesia for ovum pickup. A Second blood sample will be taken two hours after aspiration of the last follicle in recovery room post-operatively.

A third final blood sample will be taken before Embryo transfer .The blood samples will be sent immediately to central laboratory in Kasr Alainy Cairo University Hospital after being obtained on every occasion, and Serum prolactin will be analyzed by immunoassay in each time.

Descriptive data such as age, type of infertility & cause will be recorded. Also result of every serum prolactin level will be recorded as well as type of protocol used for ovulation induction, number of oocytes retrieved at ovum pick up, embryo grading and day of transfer.

Serum beta human chorionic gonadotropin (B-hCG) will be drawn from the patient 2 weeks after the date of embryo transfer to determine pregnancy and recorded.

Statistical analysis will be done for the laboratory results, All statistical calculations were performed using the computer program SPSS (Statistical Package for the Social Science; SPSS Inc.) version 15 for Microsoft Windows

.

ELIGIBILITY:
Inclusion Criteria:

* Age: adult female >20 years old.
* Complaining of infertility 1ry or 2ry & scheduled for ICSI.

Exclusion Criteria:

* Hyperprolactinemia patients.
* Severe Male factor infertility
* Frozen embryo transfer cycles
* Uterine Anomalies.
* Repeated implantation failure in ICSI.
* Any contraindications for Pregnancy as(serious uncontrolled medical diseases such as Diabetes, heart disease, hypertension), mental illnesses, ovarian tumors,cancer of any location and Acute inflammatory disease).
* On medication that is known to alter prolactin levels e.g antipsychotics, Atypical agents and risperidone
* Thyroid dysfunction.
* Medical disorders affecting serum prolactin eg acromegaly ,chronic renal failure and hypothyroidism.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ninety normo-prolactinemic patients attending the Assisted reproduction unit in the Obstetrics and Gynecology Department-Faculty of Medicine -Cairo University, Scheduled for ICSI treatment cycle .Each participant will be subjected to infertility work up investigation in the form of semen analysis, hormonal profile (FSH, LH, TSH and prolactin).
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Difference in Serum prolactin Levels (ng/mL) between ovum pickup & Embryo transfer | 6 months

SECONDARY OUTCOMES:
o Correlate serum prolactin levels (ng/mL) with Pregnancy rate. | 6 months
Correlate serum prolactin levels (ng/mL) with number & quality of embryos | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Kamel, MD, Principal Investigator — Lecturer Of obstetrics & Gynecology
Locations (1):
- 11562, Ḩadā’iq al Qubbah, Cairo Governorate, Egypt

REFERENCES:
- [Background] Boyers SP, Lavy G, Russell JB, Polan ML, DeCherney AH. Serum prolactin response to embryo transfer during human in vitro fertilization and embryo transfer. J In Vitro Fert Embryo Transf. 1987 Oct;4(5):269-72. doi: 10.1007/BF01555202. PMID 2961832
- [Derived] Kamel A, Halim AA, Shehata M, AlFarra S, El-Faissal Y, Ramadan W, Hussein AM. Changes in serum prolactin level during intracytoplasmic sperm injection, and effect on clinical pregnancy rate: a prospective observational study. BMC Pregnancy Childbirth. 2018 May 9;18(1):141. doi: 10.1186/s12884-018-1783-4. PMID 29739353